CLINICAL TRIAL: NCT06069115
Title: Investigation of Oxygen Metabolism and Reserve Capabilities of Cardiovascular and Respiratory Systems in Patients with Malignant Neoplasms of the Breast in the Course of Complex Treatment
Brief Title: Radiotherapy Exposed Lung Injury: Effect on Functioning - Cohort
Acronym: RELIEF-COHORT
Status: Recruiting | Type: Observational
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Other Study IDs: 584-н
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms; Radiation Pneumonia; Radiation Pneumonitis; Radiation Induced Fibrosis
Keywords: breast cancer; radiation therapy; radiation induced lung fibrosis
MeSH Terms: conditions — Breast Neoplasms; Radiation Pneumonitis; Radiation Fibrosis Syndrome | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main cohort group: All participants will be included in the same group, with no subgrouping within this study.
  Interventions: Radiation: Radiation therapy protocol for Breast cancer; Diagnostic Test: Spirography and assessment of pulmonary diffusion capacity; Diagnostic Test: Cardiopulmonary stress test; Diagnostic Test: Computed tomography of the chest organs; Diagnostic Test: SF-36 Quality of Life Questionnaire; Diagnostic Test: Demographic and anthropometric measures; Other: Indicators characterizing the severity of the underlying disease

INTERVENTIONS:
Radiation: Radiation therapy protocol for Breast cancer — Conformal 3D radiation therapy will be performed 4-12 weeks after surgical treatment of breast cancer on Electa Axesse linear gas pedal with 6 MeV energy in traditional fractionation mode. Different RT schemes will be used depending on the stage of the disease, type of surgical treatment, and morphological variant of the tumor. In organ-preserving surgeries the remaining breast will be irradiated with a single focal dose (FD) of 2 Gy, up to the total focal dose (TFD) of 50 Gy. In the presence of risk factors, irradiation of lymphatic outflow pathways will be performed: axillary, sub/adclavicular and parasternal lymph nodes areas (FD 2 Gy, up to TFD 44-46 Gy). In radical breast resection we'll use irradiation of the anterior chest wall in 2 Gy FD, up to 50 Gy FD, irradiation of lymphatic outflow pathways: axillary, sub/adclavicular and parasternal lymph nodes (2 Gy FD, up to 44-46 Gy FD).
Diagnostic Test: Spirography and assessment of pulmonary diffusion capacity — Using the Master Screen Body device you will be asked to take two series of breaths through a special tube for 2-3 minutes. Usually the procedure does not cause any discomfort
Diagnostic Test: Cardiopulmonary stress test — The exercise test is performed on a bicycle ergometer Oxycon Pro. Prior to the test, special sensors for recording the electrocardiogram, a sensor to determine blood saturation, and a cuff to measure blood pressure will be glued on the body. Breathing during the test takes place through a face mask with a built-in gas analyzer sensor. The stress test is conducted up to an individual maximum (according to the age, sex, height and weight of the patient), followed by a recovery period. There is some temporary discomfort associated with performing physical activity. Dyspnea, leg fatigue, and dizziness may occur. Observation continues until full recovery of hemodynamic and gas exchange parameters, in case of appearance of unfavorable symptoms - until their disappearance.
Diagnostic Test: Computed tomography of the chest organs — CT is a method of examination based on X-rays, but unlike conventional X-rays, it gives the most complete picture of the body structure, with less radiation.
  Tomography usually does not cause any unpleasant feelings and is performed in a specialized department.
  Other Names: MSCT
Diagnostic Test: SF-36 Quality of Life Questionnaire — Standard questionnaire for assessment quality of patient's life https://clinmedjournals.org/articles/jmdt/jmdt-2-023-figure-1.pdf
Diagnostic Test: Demographic and anthropometric measures — Age, sex, height. weight, body mass index (BMI)
Other: Indicators characterizing the severity of the underlying disease — Severity of underlying disease (mMRC, BODE, SMRT-CO Respiratory Support Need Scale), and comorbidities (cardiovascular disease, diabetes mellitus, chronic obstructive pulmonary disease, chronic kidney disease) Medications taken.

SUMMARY:
Prospective cohort research to study the state of oxygen metabolism, reserve capabilities of cardiovascular and respiratory systems in patients with breast cancer to create a program of prevention and rehabilitation of lung damage in the process of complex treatment of the disease.

The aim of the study is to study the dynamics of oxygen metabolism and reserve capabilities of cardiovascular and respiratory systems in the process of complex treatment of breast neoplasias.

Objectives of the study:

1. Explore the dynamics of pulmonary ventilation and gas exchange disorders in patients with breast cancer in the course of radiation therapy
2. Establish an algorithm for risk stratification of post-radiation disorders of pulmonary ventilation and gas exchange in patients with breast cancer.
3. Analyze the prognostic significance of cardiopulmonary exercise testing in assessing the cardiotoxic effect of chemo- and radiation therapy in patients with breast cancer.
4. Analyze the influence of post-radiation disorders of pulmonary ventilation and gas exchange on the quality of life and psycho-emotional status of patients with breast cancer.
5. Develop a fundamental basis for the program of prevention and rehabilitation of post-radiation lung damage in patients with breast neoplasias based on the study of individual parameters of oxygen metabolism and reserve capabilities of cardiovascular and respiratory systems.

All participants go through 5-week radiation therapy in standard protocol, will have investigation of their lung functioning by spirography and assessment of pulmonary diffusion capacity, cardiopulmonary stress tests and CT-scan on the lungs before radiotherapy course. Researchers will analyze such parameters as stage of the disease, surgery type, all patient's medications, complications, nutritional status, psychological status.

DETAILED DESCRIPTION:
After a discussion about the possibility of participating in the study, the patient is presented with an informed consent form and all questions of interest are explained. If consent to participate in the study is obtained, the patient and the researcher fill in all the required fields of two copies of the informed consent form and sign it. If necessary, the researcher re-explains any information regarding the study. One copy of the informed consent remains with the patient and the second copy is kept, as required by Good Clinical Practice, by the researcher.

Once informed consent has been obtained, an Individual Registration Card (IRC) is completed for the patient included in the study. Completion of the IRC also continues until all phases of the study are completed.

Pulmonary function tests, cardiopulmonary stress testing (CPST), indirect calorimetry are performed in patients with breast cancer who have undergone surgical treatment of the disease and referred for radiation therapy in the FGBU "NMC named after E.N. Meshalkin" of the Ministry of Health of Russia using MasterScreen Pneumo (Jaeger, Germany), Oxycon Pro ergospirometry (Jaeger, Germany), and indirect calorimetry systems for evaluation of external respiratory function in accordance with international standards. External respiration indices were adjusted to BTPS conditions (body temperature (37°C), ambient pressure and gas saturated with water vapor), and gas exchange - STPD (standard temperature (0°C or 273 K) and pressure (760 mm Hg) and no water vapor). The protocol of stress testing is selected individually, based on the proper values in accordance with the age, sex and anthropometric data of the patient. The study is conducted up to the individual maximum followed by a recovery period. The anaerobic threshold is determined using the V-slope method. After reaching the peak load, it is gradually reduced. Observation continues until full recovery of hemodynamic parameters, gas exchange, in case of adverse symptoms - until their disappearance. Repeated testing is performed in the first week after the end of the course of radiation therapy.

MSCT of the chest is performed on the 1-2 day of patient inclusion in the study to assess the initial state of the bronchopulmonary system of patients.

The SF-36 quality of life questionnaire, ECOG scale for assessing the general condition of the oncologic patient, mMRC respiratory disturbance scale, anxiety and depression scales, postcovicular functional limitations scale, and cognitive impairment scale are completed at inclusion in the study and after the course of radiation therapy.

Statistical analysis:

If the data are normally distributed, they will be compared using t-test, multivariate analysis of variance and χ2 test. If the data are not normally distributed, non-parametric tests will be used. A 95% confidence interval will be applied when calculating the mean and standard deviation/median and percentiles. Dependencies between continuous quantitative variables will be studied using linear regression, in case of discrete variables Spearman correlation will be used. Binary logistic regression will be applied to study qualitative traits having 2 categories. Manual stepwise variable inclusion technique will be used to formulate multivariate regression models with a cut-off point of significance level of 0.20. In all other cases, statistical significance will be established at a probability of type one error of less than 5%. All statistical analyses will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of malignant breast neoplasm;
* signed informed voluntary consent of the patient to participate in the study.

Exclusion Criteria:

* contraindications to the use of inhaled corticosteroids (presence of active or inactive pulmonary tuberculosis, fungal, viral or bacterial infection of the respiratory organs);
* lung diseases requiring baseline therapy with glucocorticosteroids (chronic obstructive pulmonary disease, bronchial asthma);
* mental and/or musculoskeletal impairments that make it impossible to adequately perform the exercise test, cooperate with the patient and interpret the results;
* conditions and diseases requiring emergency surgical intervention and/or observation and treatment in an ICU setting;
* patient's refusal to participate in this clinical trial at any stage of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Inborn females with all inclusion criteria are eligible
Study Population: 200 patients aged 18 years and older with established diagnosis of breast malignant neoplasm, admitted to the Federal State Budgetary Institution "Meshalkin National Medical Center" of the Ministry of Health of Russia to undergo a course of radiation therapy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-07-18 (Estimated); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2peak) | 3-6 months
  Patient's data of spirometry will be compared between values before the radiotherapy and 3 to 6 months after.

SECONDARY OUTCOMES:
Quality of life as measured by the SF-36 questionnaire. | 3-6 months
  Patient's data of questionnare will be compared between values before the radiotherapy and 3 to 6 months after.
1-year mortality from any cause | 1, 2, 3 years
  We'll contact with patient and their relatives to assess the mortality rates after radiotherapy on 1? 2 and 3 years after the treatment
Dynamics of lung diffusion capacity (∆DLCO) | 3-6 months
  Patient's data of spirometry will be compared between values before the radiotherapy and 3 to 6 months after.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana Kamenskaya, PhD, MD, Principal Investigator — Meshalkin Scientific Research Center of the Ministry of Health of Russia
Locations (1):
- Meshalkin Scientific Research Center of the Ministry of Health of Russia, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No